CLINICAL TRIAL: NCT04217694
Title: A Pilot Study Evaluating the Feasibility of Memantine in Reducing Cognitive Impairment in Pediatric Patients After Radiation Therapy for Central Nervous System Tumors
Brief Title: Memantine for the Reduction of Cognitive Impairment After Radiation Therapy in Pediatric Patients With Central Nervous System Tumors
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MC1911; NCI-2019-08538 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1911 (Other: Mayo Clinic); 19-004245 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2019-12-23; First posted 2020-01-03 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Malignant Central Nervous System Neoplasm; Primary Central Nervous System Neoplasm
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prevention (memantine, CogState) (Experimental): Patients receive memantine PO BID beginning at the time of study enrollment (no later than 1st day of RT) up to 6 months after completion of standard of care RT in the absence of unacceptable toxicity. Patients also complete CogState cognitive testing at baseline, at completion of RT, and at 3, 6, and 12 months after completion of RT.
  Interventions: Behavioral: Cogstate Assessment Battery; Drug: Memantine; Drug: Memantine Hydrochloride

INTERVENTIONS:
Behavioral: Cogstate Assessment Battery — Complete CogState testing
Drug: Memantine — Given PO
Drug: Memantine Hydrochloride — Given PO
  Other Names: Ebixia; Namenda

SUMMARY:
This early phase I trial studies the feasibility of giving memantine for the reduction of cognitive impairment after radiation therapy in pediatric patients with central nervous system tumors. Memantine may reduce the effects of radiation therapy on memory and thinking.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the feasibility of twice daily memantine started before radiation therapy (RT) and one month after RT.

SECONDARY OBJECTIVE:

I. To evaluate the feasibility of twice daily (BID) memantine started before RT and continued 3 and 6 months after RT.

EXPLORATORY OBJECTIVES:

I. To evaluate the change in neurocognitive function (NCF) as found by formal neurocognitive testing between baseline and 12 months post-RT.

II. To compare the change in NCF between baseline and the end of RT, 3,and 6 months after RT using both neuropsychological testing and the CogState exam.

III. To evaluate changes in quantitative volumetric brain imaging using Neuroquant software analysis of magnetic resonance imaging (MRI) imaging before and 12 months after radiation.

IV. To correlate cognitive changes detected by CogState composite score and formal neuropsychological testing.

V. Disease-free (of primary tumor) and overall survival.

OUTLINE:

Patients receive memantine orally (PO) BID beginning at the time of study enrollment (no later than 1st day of RT) up to 6 months after completion of standard of care RT in the absence of unacceptable toxicity. Patients also complete CogState cognitive testing at baseline, at completion of RT, and at 3, 6, and 12 months after completion of RT.

After completion of study, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Receiving intracranial radiation for a primary central nervous system (CNS) malignancy
* Histological or radiologic confirmation of intracranial disease
* Able to use the computer for CogState assessment battery
* Normal serum creatinine per institutional normal limits (obtained =< 35 days prior to study entry)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) OR direct bilirubin =< ULN for patients with total bilirubin levels > 1.5 x ULN (obtained =< 35 days prior to study entry)
* Aspartate transaminase (AST) AND alanine transaminase (ALT) =< 2.5 x ULN
* Provide informed consent if over age 18, or provide assent with consent from parent or legal guardian if age 7-17
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only. Patients capable of childbearing must use adequate contraception

Exclusion Criteria:

* Patients with World Health Organization (WHO) grade IV astrocytoma or glioblastoma tumors

  * Note: A patient with grade IV tumors of other histology can participate in the study if they meet all other criteria
* Any prior intracranial radiation
* Any contraindication or allergy to memantine
* Use of short-acting benzodiazepines (may excite lethargy/dizziness with memantine)

  * Note: occasional use as a sleep aid or as needed for anxiety or nausea is allowed
* Intractable seizures while on adequate anticonvulsant therapy, defined as more than one seizure per month for the past 2 months
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2024-08-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who attempt to take appropriate dose of memantine | At 1 month post-radiation therapy (RT)
  The rate of feasibility (the percentage of patients who attempt to take at least 80% percent of their prescribed dose) will be calculated, along with corresponding 90% confidence intervals.

SECONDARY OUTCOMES:
Percentage of patients who attempt to take appropriate dose of memantine | At 3 and 6 months post-RT
  The rate of feasibility (the percentage of patients who attempt to take at least 80% percent of their prescribed dose) will be calculated, along with corresponding 90% confidence intervals.

OTHER OUTCOMES:
Change in neurocognitive function (NCF) | Baseline up to 12 months post-RT
  Will be summarized and reported descriptively. This will be assessed using results from neurocognitive testing. Differences between scores from baseline and 12 months post-RT will be calculated, along with corresponding 90% confidence intervals. Change index (reliable change index [RCI]) will be calculated as well over this time period. A paired t-test or the Wilcoxon rank-sum test will be used as applicable. Additional analyses concerning change in NCF using additional subscales from the results of neurocognitive testing may be performed, but will be hypothesis generating and considered exploratory. These may include the use of other neurocognitive testing subscales using t-tests or the Wilcoxon rank-sum test, variations of RCI, and linear regression to assess the relationship of each subscale with changes in NCF.
Change in NCF - CogState | Baseline up to 6 months post-RT
  Determined by the CogState composite score. Will be summarized and compared to baseline values. Additional analyses concerning NCF at or between various time points may be performed, but will be hypothesis generating and considered exploratory. These may include comparisons of NCF between baseline and the end of RT, 3 months, and 12 months post-RT. Subscales of the results from the CogState may also be used for these analyses. CogState is a computerized cognitive test that will include the following battery of tests: International Shopping List Test (verbal learning and delayed recall), Detection (processing speed), Identification (attention), One Card Learning (visual memory), and One Back (working memory). Higher scores generally indicate greater NCF.
Change in NCF - neuropsychological exam | Baseline up to 6 months post-RT
  Determined by neuropsychological examination. Will be summarized and compared to baseline values. Additional analyses concerning change in NCF at or between various time points may be performed, but will be hypothesis generating and considered exploratory. These may include comparisons of NCF between baseline and the end of RT, 3 months, and 12 months post-RT .
Change in quantitative volumetric brain imaging | Baseline up to 12 months post-RT
  Neuroquant Software will be used to analyze quantitative magnetic resonance imaging measurements of changes in hippocampal volume. Differences between measurements will be reported, along with corresponding 90% confidence intervals. A paired t-test or the Wilcoxon rank-sum test will be used as applicable. Additional analyses concerning hippocampal volume may be performed, but will be hypothesis generating and considered exploratory.
Change in cognition | Baseline up to 12 months post-RT
  Cognitive changes detected by the CogState composite score will be correlated with results from formal neuropsychological testing using Pearson's r or Spearman's rank method, as applicable.
Disease-freedom from primary tumor | Up to 2 years
  Will be analyzed using Kaplan-Meier.
Overall survival | Up to 2 years
  Will be analyzed using Kaplan-Meier.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia N. Laack, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials